CLINICAL TRIAL: NCT04995302
Title: The Comparison of Microneedling Therapy With or Without Amnion Bilayer Sheeting on Post-Burn Hypertrophic Scar Tissue
Brief Title: Microneedling Therapy With or Without Amnion Bilayer Sheeting on Scar Tissue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Irma Bernadette S. Sitohang, MD, PhD - Head of Cosmetic Dermatology Division, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Organization: Indonesia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MicroneedlingScar
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Scars, Hypertrophic; Burn Scar
Keywords: Microneedling; Amnion bilayer; Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic; Cicatrix

STUDY DESIGN:
Intervention Model Description: In this study, one scar in one subject, will be divided into two areas, one-half of the scar will receive an intervention of microneedling, and the other half will receive microneedling+amnion bilayer. Hence, one subject will receive both interventions at the same time
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedling and Amnion Bilayer (Active Comparator): Microneedling is a dermaroller procedure that uses small needles to prick the skin. Amnion bilayer is used as an additional therapy after microneedling therapy.
  Interventions: Procedure: Microoneedling and Amnion Bilayer
- Microneedling (Placebo Comparator): Microneedling is a dermaroller procedure that uses small needles to prick the skin.
  Interventions: Procedure: Microoneedling

INTERVENTIONS:
Procedure: Microoneedling and Amnion Bilayer — Microneedling is conducted following a three-week application of tretinoin cream. Then, scar tissue that has been treated with microneedling is covered with amnion bilayer for 72 hours.
  Arms: Microneedling and Amnion Bilayer
Procedure: Microoneedling — Microneedling is conducted following a three-week application of tretinoin cream. Then, scar tissue that has been treated with microneedling is covered with an antibacterial gauze dressing.
  Arms: Microneedling

SUMMARY:
The aim of this study is to compare the outcome of microneedling therapy with or without amnion bilayer sheeting on post-burn hypertrophic scar tissue. A clinical trial will be conducted with 17 samples, from September to December 2021.

DETAILED DESCRIPTION:
High degree burn injuries commonly result in abnormal scar formation, and therapy for this hypertrophic scar remains a challenge. For years, microoneedling has been used for treating hypertrophic scars, and an addition of amnion bilayer sheeting is expected to provide a more favorable outcome. This study aims to compare microneedling therapy with or without amnion bilayer sheeting on post-burn hypertrophic scars tissue. This is an interventional study with 17 samples, aged 18-50 years old. Therapeutic outcomes will be evaluated using visual analog scale, degree of erythema, patient's subjective evaluation, dermoscope, biopsy, and skin ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 18-50 years old
* Patients with post-burn, mature hypertrophic scars, localized in any areas other than the face, with a minimum of 5 cm in diameter.
* Patients are willing to participate in the study and sign an informed consent form

Exclusion Criteria:

* Patients with scars less than 5 cm in diameter
* Patients with scars localized solely in the face
* Hypertrophic scars with keloid
* Patients with comorbidities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective Pain in one month | Baseline, day 7, day 30
  Using Visual Analog Scale (0-10, 0 indicates no pain and 10 indicates severe pain)
Change in Erythema Degree in one month | Baseline, day 7, day 30
  Using Erythema score (0-4, 0 indicates no erythema and 4 indicates severe erythema)
Change in Dermoscopy Evaluation in one month | Baseline, day 7 , day 30
  Qualitative description of blood vessel structure, pigmentation density and erythema
Change in Biopsy Evaluation in one month | Baseline, Day 7 and day 30
  Descriptive evaluation using HE staining
Change in Skin Thickness in one month | Baseline, Day 7 and day 30
  Evaluation with USG of epidermal and dermal layer (in pixels)
Change in Subjective Improvement in one month | Baseline , Day 7 and day 30
  Using Patient and Observer Scar Assessment Scale (Patients scored from 1-10 in pain, itch, color, stiffness, thickness and irregularity of their scar, observer gives score on vascularity, pigmentation, thickness, relief, pliability, and surface area)
Change in Subjective Improvement in one month | Baseline , Day 7 and day 30
  Using Modified Vancouver Scar Scale (Evaluating pigmentation (score 0-3), vascularity (0-3), pliability (0-5), height (0-5))

CONTACTS AND LOCATIONS:
Overall Officials: Irma B Sitohang, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- dr. Cipto Mangunkusumo Hospital, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No